CLINICAL TRIAL: NCT06107452
Title: Customization of Cardiac Readaptation Based on Force-velocity Profile and Heart Rate Variability: A Controlled and Randomized Study
Brief Title: Customization of Cardiac Readaptation Based on Force-velocity Profile and Heart Rate Variability
Acronym: PROPIU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 23CH152; 2023-A01452-43 (Other: ANSM)
Record Dates: First submitted 2023-10-11; First posted 2023-10-30 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-01

CONDITIONS: Acute Coronary Syndrome
Keywords: Cardiac rehabilitation; Physical activity; Force-velocity profile; Autonomic nervous system; Coronary artery disease
MeSH Terms: conditions — Acute Coronary Syndrome; Motor Activity; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Patient with acute coronary syndrome will be included. According to their initial strength-speed profile, coronary patients will benefit from an individualized cardiac rehabilitation program, with strength or speed training adapted to the autonomic nervous system (ANS).
  Interventions: Other: training strategy with adaptation of training strategies to the ANS
- Control group (Active Comparator): Patient with acute coronary syndrome will be included. According to their initial force-velocity profile, coronary patients will have an individualized cardiac rehabilitation program, either with a training in force or in velocity.
  Interventions: Other: training strategy (standard practice)

INTERVENTIONS:
Other: training strategy with adaptation of training strategies to the ANS — a training strategy for subjects whose PFVP is in favour of strength or speed with training load adjusted according to SNA
  Arms: Experimental group
Other: training strategy (standard practice) — a training strategy for subjects whose PFVP is in favour of strength or speed
  Arms: Control group

SUMMARY:
Cardiac readaptation aims to mitigate cardiovascular risks and enhance the quality of life among coronary patients. Our research laboratory has an international expertise in training optimization in top-athletes and a previous study has demonstrated the efficacy of optimizing cardiac rehabilitation through the power-force-velocity profile (PFVP). The findings exhibited significant improvements in aerobic capacity, muscular strength, and cardiovascular parameters among patients who were trained based on their PFVP. Guided training utilizing heart rate variability (HRV) is also garnering increasing interest as a means to optimize training load and promote recovery

DETAILED DESCRIPTION:
Our study aims to evaluate the application of HRV in regulating training load based on fatigue levels in cardiac rehabilitation patients utilizing the PFVP framework.

ELIGIBILITY:
Inclusion Criteria:

* >18
* Acute Coronary Syndrome treated in the last 6 months
* Medical revascularization (angioplasty ± stenting) or surgical (coronary artery bypass)
* Initial CPETt: MPA ≥ 60w in women and ≥80w in men
* French
* Informed consent

Exclusion Criteria:

- Significant co-morbidities limited practice of physical activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
The root mean square of successive differences in heart rate or RMSSD | Baseline to 2 months
  The root mean square of successive differences in heart rate or RMSSD will be measured from a nocturnal Holter ECG recording at the end of 8 weeks of exercise retraining and compared with the initial pre-training value. weeks of exercise re-training and compared with the initial pre-training value.

SECONDARY OUTCOMES:
Value of maximum oxygen consumption | Baseline to 2 months
  VO2 max (ml/min/kg) thanks to 24-hour ECG recording
Assessment of the ANS sympathetic branch | Baseline to 2 months
  Assessment of the ANS sympathetic branch thanks to SDNN index value
Assessment of the ANS parasympathetic branch | Baseline to 2 months
  Assessment of the ANS parasympathetic branch thanks to RMSSSD index value
non-invasive measurement of arterial stiffness | Baseline to 2 months
  value of pulse wave propagation velocity
measurement of upper and lower limb muscle strength | Baseline to 2 months
  it's a composite outcome :
  * measurement of handgrip (kg) thanks to Jamar hydraulic hand dynamometer
  * measurement maximum quadriceps strength (kg) thanks to Contrex, Physiomed
assessment of PFVP evolution | Baseline to 2 months
  assessment of PFVP evolution thaks to cycloergometer sprint (Monark, Vansbro)
assessment of physical a activity and sedentary behavior | Baseline to 2 months
  it's a composite outcome :
  * assessment of physical a activity and sedentary behavior thanks to actimetry (Actigraph GT9x)
  * assessment of physical a activity and sedentary behavior thanks to Adult Physical Activity Questionnaire (APAQ)
quality of life assessment | Baseline to 2 months
  it's a composite outcome :
  * with mental quality of life score
  * with physical quality of life score
assessment of subjective fatigue | Baseline to 2 months
  assessment of subjective fatigue thanks to FACIT-F questionary
biological data | Baseline to 2 months
  it's a composite outcome : complete blood biology and relevant inflammatory biomarkers involved in cardiac rehabilitation.

CONTACTS AND LOCATIONS:
Overall Officials: David HUPIN, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No